CLINICAL TRIAL: NCT05362474
Title: Targeting Leukotrienes in Kidney Disease: A Pilot Study
Brief Title: Targeting Leukotrienes in Kidney Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not available
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0187
Record Dates: First submitted 2022-04-21; First posted 2022-05-05 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- montelukast (Experimental): montelukast 10mg orally once a day
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — 10mg orally once a day

SUMMARY:
Diabetic kidney disease (DKD) is associated with significant morbidity and mortality. Identifying new treatments for DKD to be used alone or in combination with other therapies is a high priority. Inflammation plays a key role in DKD and targeting pro-inflammatory lipid mediators called leukotrienes may represent a promising therapy for DKD. The current proposal will investigate whether montelukast, a leukotriene antagonist, reduces proteinuria and improves vascular function and arterial stiffness in patients with DKD.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 3
* urine albumin to creatinine ratio 200-5000 mg/g
* blood pressure <140/90 mmHg
* use of angiotensin converting enzyme inhibitor or angiotensin receptor blocker with stable dose for 4 weeks
* history of diabetes type 1 or 2
* BMI <40 kg/m2
* Stable antihypertensive regimen for at least one month prior to enrollment
* Stable diabetes regimen for at least one month prior to enrollment
* Sedentary or recreationally active (<2 days of vigorous aerobic exercise as vigorous exercise may affect vascular function measurements)
* Able to provide consent

Exclusion Criteria:

* Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Uncontrolled hypertension
* Factors judged to limit adherence to interventions (e.g. history of medication noncompliance, noncompliance with follow up visits, significant cognitive impairment, etc.)
* Anticipated initiation of dialysis or kidney transplantation within 3 months
* Current participation in another research study
* Pregnancy or planning to become pregnant or currently breastfeeding
* Allergy to aspirin
* Severe hepatic impairment (Child-Pugh Class C)
* History of major psychiatric disorder
* Use of inhaled or systemic corticosteroids or long-acting beta agonists (higher risk of neuropsychiatric reaction)
* Current use of SGLT2 inhibitor
* Current use of phenobarbital, rifampin or carbamazepine.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Montelukast
Started | 6
Completed (5) | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Montelukast
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Albuminuria at 3 Months
Description: Change in 24-hour urine albumin excretion at 3 months
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Montelukast
Number analyzed (Participants) | 5
mg/day
  Baseline | 1.84 (1.96)
  3 months | 1.05 (0.44)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Montelukast
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05362474/Prot_SAP_001.pdf